CLINICAL TRIAL: NCT02146885
Title: The Use of Diffuse Optical Spectroscopy to Characterize Adipose Tissue Oxygenation and Vascular Reactivity in Response to Weight-Loss Intervention
Brief Title: The Use of Diffuse Optical Spectroscopy to Characterize in Response to Weight-Loss Intervention
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Shaista Malik, M.D., Assistant Professor-Cardiology, University of California, Irvine
Other Study IDs: 20129158
Record Dates: First submitted 2014-05-19; First posted 2014-05-26 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Weight Control: Weight Control
  Interventions: Other: Weight Control

INTERVENTIONS:
Other: Weight Control — Weight Control

SUMMARY:
The first step in any clinical intervention against obesity involves sustained lifestyle changes. Researcher can use these strategies to beneficial the effects of weight and on cardiovascular risk. The researcher develope methods for assessing the effectiveness use optical technology to make such assessments, specifically in the area of fatty tissue can predict the effectiveness of the intervention in causing weight reduction and treating metabolic disease.

DETAILED DESCRIPTION:
Optical technologies under development at the Beckman Laser Institute.

Diffuse Optical Spectroscopy Imaging is a method for studying absorption and scattering (optical properties) of tissue in humans. It is related to near-infrared spectroscopy , but allows for more quantitative and thorough measurements. The researcher use Diffuse Optical Spectroscopy to measure fatty tissue, water, blood concentration level during weight loss program to determine the effect of sustained changes in weight or relapses.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index greater than 25, overweight
* Participation in Weight Loss program

Exclusion Criteria:

* A medical history of myocardial infarction or cerebrovascular stroke
* Pregnancy or planned pregnancy during the course of the study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population will be selected from University of California Irvine Medical Center Department of Cardiology, preventive cardiology intervention program.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2013-01-08 (Actual); Primary Completion 2017-01-13 (Actual); Study Completion 2017-01-13 (Actual)

PRIMARY OUTCOMES:
Weight Control | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Shaista Malik, MD, Principal Investigator — Beckman Laser Institute, UCI
Locations (1):
- Beckman Laser Institute, Irvine, California, United States